CLINICAL TRIAL: NCT01304940
Title: The Psychophysiology and Neurobiology of PTSD Across the Menstrual Cycle
Brief Title: Women's Post Traumatic Stress Disorder (PTSD) Research Study
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Boston VA Research Institute, Inc. (Other); Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: CDA-2-042-07F
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, blood and saliva samples are taken. Only blood and saliva samples are retained and used to measure stress hormone levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PTSD group: Individuals in this group meet criteria for PTSD as defined by DSM-IV
- trauma control group: individuals in this group do not meet criteria for any Axis I diagnosis as defined by DSM-IV

SUMMARY:
The purpose of this study is to examine the relationship between trauma and startle. The investigators are also looking at the effect of menstrual phase on this relationship.

DETAILED DESCRIPTION:
The investigators are trying to understand if there is a relationship between the experience of traumatic events such as those experienced by people with post traumatic stress disorder and reactivity to startling noises or mild threats. So, the investigators are looking at startle reflex, heart rate, and stress hormone responses to short noises and small shocks in people exposed to trauma and who either do or do not have PTSD. Additionally, the investigators will be looking at how the menstrual cycle impacts these processes. The investigators know that women have twice the risk for developing PTSD and some research suggests that stress hormones change during the menstrual cycle and may have an effect on risk.

ELIGIBILITY:
Inclusion Criteria:

* Women, ages 18-55 years old who have a regular menstrual cycle and who can come in to participate in the afternoon

Exclusion Criteria:

* Long-term medications, oral or steroid contraceptives, irregular menstrual cycle

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women, ages 18-55.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2013-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Pineles, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTSD Group | Trauma Control Group
Started | 25 | 25
Completed Study | 25 (recruitment ended when 25 participants completed study procedures) | 25 (recruitment ended when 25 participants completed study procedures)
Completed | 22 (these participants met severity requirement and were included in study analyses) | 25
Not Completed | 3 | 0
Not completed — not meet symptom severity requirement | 3 | 0

BASELINE CHARACTERISTICS:
Population: Additional PTSD subjects were dropped from analyses due to low severity
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Group | Trauma Control Group | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 20 | 25 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 5 | 10 | 15
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 25 | 47
smokers [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Prepulse Inhibition
Description: To calculate prepulse inhibition (PPI), first an O-EMG response score (O-EMG-R) for each trial was calculated. O-EMGR was measured in microvolts and each value was subjected to a square root transformation. For each participant, the mean O-EMG-R scores were calculated for both startle alone and prepulse + startle trials across the entire session. PPI is a ratio and was calculated by the formula below:
  PPI=(mean OEMG-R score on prepulse+startle trials-mean OEMG-R on Startle alone trials)/mean OEMG-R on startle alone trials.
  A negative value on this PPI ratio is indicative of greater prepulse inhibition.
  Means and SEs below reflect estimated means and SEs for the PTSD group and trauma control group from the ANOVA conducted with menstrual phase and the PTSD group X menstrual phase interaction included in the model.
Time Frame: This measure was assessed twice for each participant, once in the midluteal phase of the menstrual cycle and once in the early follicular phase of the menstrual cycle, up to approximately 20 days apart.
Population: all participants with valid psychophys data analyzed
Measure: Mean (Standard Error); unit: proportion of change in OEMGR response
Arm/Group | PTSD Group | Trauma Control Group
Number analyzed (Participants) | 22 | 25
proportion of change in OEMGR response | -.19 (.04) | -.31 (.04)

ADVERSE EVENTS:
Arm/Group | PTSD Group | Trauma Control Group
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes